CLINICAL TRIAL: NCT01686932
Title: Multicentric Cross-over Trial to Assess the Glycemic Profiles on 8 Weeks of Vildagliptin and Sitagliptin Treatment, Each, in Type-2 Diabetic Patients With a Pre-existing Cardiovascular Disease Pre-treated With Insulin, Using a PROBE-design
Brief Title: Vildagliptin vs Sitagliptin add-on to Insulin - Impact on Glycemic Profile and Correlation of Hypoglycemic Episodes and Heart Function
Acronym: CGM-VISIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ADE07
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: vildagliptin; sitagliptin; continuous glucose monitoring (CGM); glycemic fluctuations; MAGE; impact of hypoglycemia on heart function (cardiac dysfuction measured via ECG); difference in glycemic profile of vildagliptin compared to sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin followed by Sitagliptin (Experimental): Period 1: vildagliptin 50mg BID for 8 weeks; followed by Washout then Period 2: sitagliptin 100mg QD for 8 weeks
  Interventions: Drug: Vildagliptin; Drug: Sitagliptin
- Sitagliptin followed by Vildagliptin (Experimental): Period 1: sitagliptin 100mg QD for 8 weeks; followed by Washout then Period 2: vildagliptin 50mg BID for 8 weeks
  Interventions: Drug: Vildagliptin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Vildagliptin — vildagliptin 50mg BID for 8 weeks
  Other Names: Vildagliptin (Galvus) LAF237
Drug: Sitagliptin — sitagliptin 100mg QD for 8 weeks
  Other Names: sitagliptin, Januvia

SUMMARY:
Vildagliptin and Sitagliptin both belong to the class of DPP-4 inhibitors, but differ in their pharmacokinetic profile as well as in their approved application (Vildagliptin, 2x 50 mg daily, Sitagliptin, 1x 100 mg daily). This leads to distinct results regarding postprandial blood-glucose normalization as well as protective properties regarding hypoglycemic episodes - especially during the night. Additionally, in type 1 diabetic patients a correlation has been described between hypoglycemia and abnormal heart function (QTc-elongation), which can have severe consequences for the patients. This study aims for the evaluation of the potency of both drugs to prevent and/or reduce hypoglycemic events in insulin-dependent type-2 diabetics and furthermore to evaluate the correlation of hypoglycemic episodes with changes in heart-function measured by Holter-ECG.

The hypothesis is tested, if vildagliptin leads to a more favourable glycemic profile than sitagliptin and is more potent in protecting from nocturnal abnormalities in heart-function caused by undetected hypoglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent must be obtained before any assessment is performed.

  2. Ability to comply with all study requirements. 3. Patients with Type 2 diabetes treated with stable, once or twice daily doses (minimal dose of 0.3 unit/kg/day) of basal long-acting or intermediate-acting insulin alone or in pre-mixed combination with rapid-acting or short-acting insulin for at least 12 weeks prior to Visit 1. Stable is defined as ±10% of the Visit 1 dose during the previous 12 weeks.

  4. Patients receiving metformin must be on a stable dose of metformin (at least 1500 mg daily or a maximally tolerated dose) for at least 12 weeks prior to Visit 1. 5. HbA1c ≥7.5 to ≤ 9,0% at Visit 1 6. Known CV disease based on a documented history of one or more of pre-defined criteria 7. Age: ≥40 to ≤80 years at Visit 1

Exclusion Criteria:

* 1. FPG ≥ 270 mg/dL (15 mmol/L) at Visit 1. 2. Use of any of the following medications as assessed at Visit 1:

  1. rapid or short acting insulin except in pre-mixed formulations with intermediate or long-acting insulin; insulin administration more frequently than twice-daily, or total insulin dose < 0.3 unit/kg/day for the past 12 weeks
  2. use of any oral antidiabetic medication or GLP-1 analogues within the last 12 weeks, except metformin
  3. use of weight control products including weight-loss medications in the last 12 weeks.
  4. use of oral (≥7 consecutive days) or chronic parenteral or intra-articular corticosteroid treatment within the last 8 weeks. Inhaled or topical steroids without systemic effects will be allowed.
  5. treatment with growth hormone within the previous 6 months.
  6. treatment with any drug of known and frequent toxicity to a major organ, or that may interfere with the interpretation of the efficacy and safety data during the study.

     3. a history or evidence of any of the following at Visit 1:

  <!-- -->

  1. acute metabolic conditions such a ketoacidosis, lactic acidosis or hyperosmolar state (including precoma and coma) within the past 6 months.
  2. current diagnosis of congestive heart failure (NYHA III or IV).
  3. myocardial infarction within the past 6 months.
  4. coronary artery bypass surgery or percutaneous coronary intervention within the past 6 months.
  5. Stroke, transient ischemic attack, or reversible ischemic neurologic deficit within the past 6 months.
  6. unstable angina within the past 6 months.
  7. sustained and clinically relevant ventricular arrhythmia (patients with premature ventricular contractions if deemed not clinically significant may be enrolled).
  8. Patients with permanent atrial fibrillation or pacemaker.
  9. active substance abuse, alcohol abuse and history of alcohol-related diseases within the past 2 years.
  10. type 1 diabetes, monogenic diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes (e.g. Cushing's syndrome or acromegaly-associated diabetes).
  11. malignancy of an organ system (other than localized basal cell carcinoma of the skin) treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
  12. hepatic disorder defined as:

      * acute or chronic liver disease, evidence of hepatitis, cirrhosis or portal hypertension.
      * history of imaging abnormalities that suggest liver disease (except hepatic steatosis), such as portal hypertension, capsule scalloping, cirrhosis.
  13. acute infections which may affect blood glucose control within the past 4 weeks.

      4. any of the following significant laboratory abnormalities as assessed at Visit 1:

  <!-- -->

  1. clinically significant increase or reduction in thyroid stimulating hormone (TSH) outside of the normal range.
  2. clinically significant renal dysfunction: glomerular filtration rate (GFR) <50 mL/min/1.73m2 (via MDRD formula).
  3. Patients on metformin with a GFR <60 mL/min/1.73m2 (via MDRD formula).
  4. alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN) at Visit 1, confirmed by repeated measurements within 3 working days.
  5. total bilirubin > 2 x ULN and/or direct bilirubin > 1 x ULN confirmed by repeated measurements within 3 working days.
  6. positive Hepatitis B surface antigen (HBsAg).
  7. positive Hepatitis C virus (HCV) antibody test (anti-HCV).
  8. elevated fasting triglycerides (TGs) > 500mg/dL (5.65mmol/L), confirmed by a repeated measurements within 3 working days.
  9. clinically significant laboratory abnormalities which, in the opinion of the investigator, cause the patient to be considered inappropriate for inclusion in the study.

     5. any of the following electrocardiographic abnormalities at Visit 1:

  <!-- -->

  1. second or third degree atrio-ventricular block.
  2. A QTc of > 440 ms.
  3. clinically significant electrocardiogram (ECG) abnormalities which, in the opinion of the investigator, may cause the patient to be considered inappropriate for inclusion in the study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Sulzbach-Rosenberg
  - Novartis Investigative Site, Wallerfing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period 1: 8 weeks treatment with vildagliptin 50mg BID or sitagliptin 100mg QD, 1-4 weeks wash-out, followed by Period 2, 8 weeks treatment with sitagliptin 100mg QD or vildagliptin 50mg BID
Period: Period 1
Arm/Group | Vildagliptin Followed by Sitagliptin | Sitagliptin Followed by Vildagliptin
Started | 25 | 26
Completed | 24 | 25
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Period 2
Arm/Group | Vildagliptin Followed by Sitagliptin | Sitagliptin Followed by Vildagliptin
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin Followed by Sitagliptin | Sitagliptin Followed by Vildagliptin | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.0) | 65.2 (8.6) | 65 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Profile of Vildagliptin Compared to Sitagliptin Over 4 Days After 8 Weeks of Treatment in Period 1 & 2
Description: The hypoglycemic profile is defined as the area under the curve glucose-time profile obtained by continuous glucose monitoring Interstitial glucose values below 3.9 mmol/L (averaged over 5 minutes) were considered relevant for the estimation of the interstitial glucose AUC in the hypoglycemic range These AUC<3.9mmol/L/5min. values were summed up over 4 days (unit: mmol/L/4d) or over 24 hours at measurement Days 2, 3, 4, and 5 (unit: mmol/L/24h). Lower values for AUC reflect less intense hypoglycemia.
Time Frame: baseline and 0-24 hours post-dose on Days 2 to 5
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: mmol/L/4d
Groups:
- Vitagliptin: For all Vitagliptin 50mg BID for 8 weeks in Period 1 and 8 weeks in Period 2
- Sitagliptin: For all Sitagliptin 100mg QD for 8 weeks in Period 1 and 8 weeks in Period 2
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
mmol/L/4d | 11.2 (25.65) | 5.3 (11.70)

2. Secondary Outcome: Number of Hypoglycemic Events During Vildagliptin Treatment Compared to Sitagliptin Treatment.
Description: Hypoglycemic events are defined as blood glucose values <70 mg/dL measured by a self-monitored blood glucose (SMBG) or continuous glucose monitoring (CGM) measurement regardless of any symptoms suggestive of low blood glucose.
Time Frame: after 8 weeks period 1 and Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Number; unit: number of hypoglycemic events
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
number of hypoglycemic events
  continuous glucose monitoring (CGM) | 69 | 37
  self-monitored blood glucose (SMBG) | 29 | 13

3. Secondary Outcome: Mean Duration of Hypoglycemic Events (Min.) Measured With Continuous Glucose Monitoring (CGM) Over 4 Days After 8 Weeks of Treatment for Period 1 & Period 2
Description: the mean duration of hypoglycemic events is detected by continuous glucose monitoring (CGM)measurement.
Time Frame: after 8 weeks for Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
minutes | 29.1 (44.71) | 28.0 (51.45)

4. Secondary Outcome: Mean Amplitudes of Hypoglycemic Events (mmol/L) Measured With Continuous Glucose Monitoring (CGM) Over 4 Days After 8 Weeks of Treatment for Period 1 & Period 2
Description: To evaluate by CGM measurement the grade of severity of hypoglycemia measured as the mean amplitude over 4 days after 8 weeks of treatment in Period 1 & Period 2
Time Frame: after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
mmol/L | 0.2 (0.32) | 0.2 (0.36)

5. Secondary Outcome: Number of Severe Hypoglycemic Events During Vildagliptin Treatment Compared to Sitagliptin Treatment After 8 Weeks of Treatment in Period 1 and Period 2
Description: Severe hypoglycemic events are defined as any episode requiring the assistance of another party or measured plasma glucose levels of <40 mg /dL. Assessed by self-monitored blood glucose (SMBG)After 8 weeks of treatment in Period 1 and Period 2
Time Frame: after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Number; unit: severe hypoglycemic events
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
severe hypoglycemic events | 1 | 1

6. Secondary Outcome: Glucose Fluctuations During the Day Under Vildagliptin Treatment Compared to Sitagliptin Treatment on Day 2 After 8 Weeks of Treatment Period 1 & Period 2
Description: Glucose fluctuations are assessed by the mean amplitude of glycemic excursions (MAGE) and standard deviations (SD) (Service et al., 1970). on day 2 after 8 weeks of treatment Period 1 & Period 2
Time Frame: Day 2 after 8 weeks of treatment Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
mmol/L | 4.7 (1.69) | 4.6 (1.36)

7. Secondary Outcome: Number of Participants With ECG Abnormalities Depending on Hypoglycemic Events After 8 Weeks of Treatment Period 1 & Period 2
Description: ECG abnormalities are defined as either: • Occurrence of >30 ventricular extrasystoles (VES) per hour or • Occurrence of ≥2 consecutive VES (Couplets) or • Occurrence of ≥3 consecutive VES (Triplets) or • QT-time corrected for heart rate (QTc) >440 ms. after 8 weeks of treatment Period 1 & Period 2
Time Frame: after 8 weeks of treatment Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Number; unit: participants
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
participants
  Patients with hypoglycemia (n=21,17) | 14 | 10
  Patients without hypoglycemia (n=28,32) | 19 | 24

8. Secondary Outcome: Change From Baseline of Inflammatory Biomarkers High Sensitivity C-reactive Protein (hsCRP) After 8 Weeks of Treatment in Period 1 & Period 2
Description: The inflammatory biomarkers hsCRP was assessed at baseline and after 8 weeks of treatment Period 1 & Period 2
Time Frame: Baseline, after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
mg/L | 0.79 (4.96) | 0.60 (2.48)

9. Secondary Outcome: Change From Baseline of Inflammatory Biomarkers Interleukin 6 (IL-6) After 8 Weeks of Treatment in Period 1 & Period 2
Description: The inflammatory biomarkers IL-6 was assessed at baseline and after 8 weeks of treatment Period 1 & Period 2
Time Frame: Baseline, after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: pg/L
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
pg/L | 0.40 (3.90) | 0.08 (0.93)

10. Secondary Outcome: Percentage Change From Baseline of Pro-insulin/C-peptide Ratios After 8 Weeks of Treatment Period 1 & Period 2
Description: Percentage Change from baseline of pro-insulin/C-peptide ratios after 8 weeks of treatment Period 1 & Period 2 Higher pro-insulin / C-peptide ratios (expressing disproportional hyperproinsulinemia) may be associated with increasing beta cell dysfunction and more inefficient pro-insulin processing
Time Frame: Baseline, after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
Percentage Change | -0.34 (0.47) | -0.31 (0.57)

11. Secondary Outcome: Number of Occurrence of Pre-defined ECG Findings During 4 Days of Continuous ECG Monitoring at Baseline and in the 8th Week of Periods 1 and 2
Description: Number of Occurrence of pre-defined ECG findings during 4 days of continuous ECG monitoring at baseline and in the 8th week of Periods 1 and 2. ECG data were continuously recorded and analyzed over a period of 4 days simultaneously with continuous glucose monitoring. It assessed number of any Vertical Electric(al) Sounding (VES), number of 2 consecutive VES [couplets], and number of >3 consecutive VES [salves]
Time Frame: after 8 weeks Period 1 & Period 2
Population: Full Analysis Set (FAS) included all patients that was treated with study medication.
Measure: Mean (Standard Deviation); unit: number of occurrence
Arm/Group | Vitagliptin | Sitagliptin
Number analyzed (Participants) | 49 | 49
number of occurrence
  # any VES Per.1 n=23, 25 | 879.7 (1405.2) | 2786.7 (6507.7)
  # any VES Per.2 n=25, 23 | 4389.9 (16692) | 1060.2 (1812.4)
  # couplets VES Per.1 n=23, 25 | 12.8 (32.5) | 115.0 (405.9)
  # couplets VES Per.2 n=25, 23 | 6.7 (10.3) | 2.4 (3.0)
  # salves VES Per.1 n=23, 25 | 1.0 (2.4) | 15.8 (52.6)
  # salves VES Per.2 n=25, 23 | 0.8 (1.7) | 0.9 (1.9)

ADVERSE EVENTS:
Groups:
- Vildagliptin: For all Vitagliptin 50mg BID for 8 weeks in Period 1 and 8 weeks in Period 2
Arm/Group | Vildagliptin | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 2/50 | 1/50
Other Adverse Events (participants affected / at risk) | 16/50 | 9/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin (N=50) | Sitagliptin (N=50)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin (N=50) | Sitagliptin (N=50)
BLOOD GLUCOSE DECREASED (Investigations) | 4 | 3
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.